CLINICAL TRIAL: NCT07195799
Title: A Multicenter Prospective Study of Linperlisib Combination With Cyclophosphamide, Prednisone, and Thalidomide (CPT) in Relapsed and/or Refractory Non-Hodgkin Lymphoma
Brief Title: Linperlisib Combination With Cyclophosphamide, Prednisone, and Thalidomide (CPT) in R/R NHL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-SR-219
Record Dates: First submitted 2024-11-12; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2024-12

CONDITIONS: Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- PTCL (Experimental)
  Interventions: Drug: Linperlisib combined with CPT regimen
- NK/TCL (Experimental)
  Interventions: Drug: Linperlisib combined with CPT regimen
- CLL (Experimental)
  Interventions: Drug: Linperlisib combined with CPT regimen
- MZL (Experimental)
  Interventions: Drug: Linperlisib combined with CPT regimen
- MCL (Experimental)
  Interventions: Drug: Linperlisib combined with CPT regimen
- FL (Experimental)
  Interventions: Drug: Linperlisib combined with CPT regimen

INTERVENTIONS:
Drug: Linperlisib combined with CPT regimen — Linperlisib: 80mg QD during the cycle 1-2，80mg QD for the first 7 days of cycle 3-6 (each cycle is 28 days) Cyclophosphamide: 50mg QD during the cycle 1-6 (each cycle is 28 days) Prednisone: 20mg QD during the cycle 1-6 (each cycle is 28 days) Thalidomide: 50mg QD during the cycle 1-6 (each cycle is 28 days) After six cycles, patients with CR or PR continue to receive linperlisib at a dose of 80mg for the first 7 days every cycle (each cycle is 28 days) until disease progression, intolerable toxicity, investigator judgment that treatment should be discontinued, or subject withdrawal of consent, whichever occurred first.
  Arms: CLL
Drug: Linperlisib combined with CPT regimen — Linperlisib: 80mg QD during the cycle 1-2，80mg QD for the first 7 days of cycle 3-6 (each cycle is 28 days) Cyclophosphamide: 50mg QD during the cycle 1-6 (each cycle is 28 days) Prednisone: 20mg QD during the cycle 1-6 (each cycle is 28 days) Thalidomide: 50mg QD during the cycle 1-6 (each cycle is 28 days) After six cycles, patients with CR or PR continue to receive linperlisib at a dose of 80mg for the first 7 days every cycle (each cycle is 28 days) until disease progression, intolerable toxicity, investigator judgment that treatment should be discontinued, or subject withdrawal of consent, whichever occurred first.
  Arms: FL
Drug: Linperlisib combined with CPT regimen — Linperlisib: 80mg QD during the cycle 1-2，80mg QD for the first 7 days of cycle 3-6 (each cycle is 28 days) Cyclophosphamide: 50mg QD during the cycle 1-6 (each cycle is 28 days) Prednisone: 20mg QD during the cycle 1-6 (each cycle is 28 days) Thalidomide: 50mg QD during the cycle 1-6 (each cycle is 28 days) After six cycles, patients with CR or PR continue to receive linperlisib at a dose of 80mg for the first 7 days every cycle (each cycle is 28 days) until disease progression, intolerable toxicity, investigator judgment that treatment should be discontinued, or subject withdrawal of consent, whichever occurred first.
  Arms: MCL
Drug: Linperlisib combined with CPT regimen — Linperlisib: 80mg QD during the cycle 1-2，80mg QD for the first 7 days of cycle 3-6 (each cycle is 28 days) Cyclophosphamide: 50mg QD during the cycle 1-6 (each cycle is 28 days) Prednisone: 20mg QD during the cycle 1-6 (each cycle is 28 days) Thalidomide: 50mg QD during the cycle 1-6 (each cycle is 28 days) After six cycles, patients with CR or PR continue to receive linperlisib at a dose of 80mg for the first 7 days every cycle (each cycle is 28 days) until disease progression, intolerable toxicity, investigator judgment that treatment should be discontinued, or subject withdrawal of consent, whichever occurred first.
  Arms: MZL
Drug: Linperlisib combined with CPT regimen — Linperlisib: 80mg QD during the cycle 1-2，80mg QD for the first 7 days of cycle 3-6 (each cycle is 28 days) Cyclophosphamide: 50mg QD during the cycle 1-6 (each cycle is 28 days) Prednisone: 20mg QD during the cycle 1-6 (each cycle is 28 days) Thalidomide: 50mg QD during the cycle 1-6 (each cycle is 28 days) After six cycles, patients with CR or PR continue to receive linperlisib at a dose of 80mg for the first 7 days every cycle (each cycle is 28 days) until disease progression, intolerable toxicity, investigator judgment that treatment should be discontinued, or subject withdrawal of consent, whichever occurred first.
  Arms: NK/TCL
Drug: Linperlisib combined with CPT regimen — Linperlisib: 80mg QD during the cycle 1-2，80mg QD for the first 7 days of cycle 3-6 (each cycle is 28 days) Cyclophosphamide: 50mg QD during the cycle 1-6 (each cycle is 28 days) Prednisone: 20mg QD during the cycle 1-6 (each cycle is 28 days) Thalidomide: 50mg QD during the cycle 1-6 (each cycle is 28 days) After six cycles, patients with CR or PR continue to receive linperlisib at a dose of 80mg for the first 7 days every cycle (each cycle is 28 days) until disease progression, intolerable toxicity, investigator judgment that treatment should be discontinued, or subject withdrawal of consent, whichever occurred first.
  Arms: PTCL

SUMMARY:
This is a multicenter, open-label, non-randomized, multi-cohort study to evaluate the efficacy and safety of linperlisib combined with cyclophosphamide, prednisone, and thalidomide (CPT) regimen in the treatment of relapsed and/or refractory non-Hodgkin lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, ≥18 years old;
2. Histologically confirmed diagnosis of FL/PTCL/NKTCL/CLL /MZL/MCL;
3. Except for CLL (using the 2018 iwCLL criteria), patients must have at least one measurable lesion/evaluable lesion that meets the 2014 version of Lugano lymphoma evaluation criteria;
4. FL patients:

Should be relapsed after second-line or more systemic therapy (CD20 monoclonal antibody and at least one alkylating agent, including but not limited to bendamustine, fludarabine, cyclophosphamide, isocyclophosphamide, etc.); 5. PTCL patients:

1. Have previously received at least one-line systemic treatment, have disease progression during or after the most recent treatment, or confirmed no objective response with adequate treatment;
2. Includes the following subtypes: PTCL-NOS, AITL, ALK+ALCL, ALK-ALCL，EATL; patients with ALCL must have previously received CD30-targeted therapy or be ineligible for CD30-targeted therapy; 6. NK/TCL patients:

1) Have previously received at least one line systemic treatment, have disease progression during or after the most recent treatment, or have confirmed no objective response with adequate treatment; 2) Have previously received a regimen containing Pegaspargase or L-Pegaspargase; 7. CLL patients:

1. Have measurable lesions (peripheral blood B lymphocytes ≥5×10^9/L, or enlarged lymph node (baseline LDi ≥ 1.5cm), or hepatomegaly or splenomegaly due to CLL);
2. Patients with resistance or intolerance following prior first-line or above therapy (regiments containing BTK inhibitors or BCL-2 inhibitors);
3. Treatment should be initiated when at least one indication for treatment according to IWCLL guideline are present; 8. MZL patients: Should have previously received at least two-line systemic therapy containing CD20 monoclonal antibodies and have not achieved at least partial response (PR) after recent systemic therapy, or have confirmed disease progression after treatment, and investigators judge that effective and standard treatment options are lacking; 9. MCL patients:

Previous second-line or higher treatment regimen including:

1. at least first-line immunotherapy or chemical immunotherapy containing anti-CD20 monoclonal antibody; Or anti-CD20 mab combined with BTK inhibitors;
2. have been treated with at least one appropriate BTK inhibitor and BCL-2 inhibitor (monotherapy or in combination with other antineoplastic agents); 10. ECOG PS: 0~2; 11. Expected survival ≥ 3 months; 12. Good organ function; 13. The washout period from the end of any previous antineoplastic therapy, including radiation therapy, chemotherapy, hormone therapy, surgery, or molecular-targeted therapy until participate in the trial should be at least 28 days or five half-life of the drug, whichever was shorter; 14. Fertile male and female subjects are willing to use effective contraceptive measures throughout the study period and for six months after the last dose; 15. Volunteer to participate in clinical studies and sign informed consent, willing to follow and able to complete all trial procedures.

Exclusion Criteria:

Patients with any of the following conditions are not eligible to participate in this study:

1. Had been progressed on PI3K inhibitor before enrollment;
2. Any other anti-tumor therapy within 4 weeks;
3. The presence of third-space effusion (e.g., massive pleural effusion and ascites) that could not be controlled by drainage or other methods;
4. Involvement of the central nervous system (meninges or brain parenchyma);
5. Long-term use of corticosteroids exceeding 30mg/day of prednisone or its equivalent;
6. Inability to swallow, chronic diarrhea or intestinal obstruction, or other factors affecting drug intake and absorption;
7. Individuals with a history of allergies or known hypersensitivity to any component of the regimen;
8. A history of any cardiac disease, including: (1) angina; (2) arrhythmias requiring clinical intervention; (3) myocardial infarction; (4) heart failure; (5) any other cardiac conditions deemed unsuitable for participation in this trial by the investigator;
9. Active viral, bacterial, or fungal infections requiring treatment (such as pneumonia);
10. Uncontrolled diabetes, pulmonary fibrosis, acute lung disease, interstitial lung disease, or liver failure;
11. Individuals with HBV or HCV infection (defined as positive for HbsAg and/or HbcAb with detectable HBV DNA copies) or positive for active hepatitis C (HCV) antibodies;
12. A history of immunodeficiency, including positive HIV testing, or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation, or a history of allogeneic bone marrow or hematopoietic stem cell transplantation;
13. Received autologous hematopoietic stem cell transplantation within 90 days prior to the first dose of study treatment;
14. Could not receive preventive treatment for pneumocystis, HSV, or HZV at screening;
15. Major surgery within 2 weeks before starting treatment;
16. Any adverse event related to prior treatment, but has not recovered to grade ≤ 1;
17. Existing active bleeding or new thrombotic disease, or have a history of bleeding tendency;
18. Pregnant or breastfeeding female patients, or women of childbearing potential with a positive baseline pregnancy test;
19. Concomitant diseases (such as severe hypertension, diabetes, thyroid disease, etc.);
20. Other malignancies within the last 5 years, except cured basal cell carcinoma of the skin and carcinoma in situ of the cervix;
21. Received live attenuated vaccines within 30 days prior to the first dose;
22. Histologically or cytologically confirmed patients with grade 3b follicular lymphoma, and known follicular lymphoma transformed into diffuse large B-cell lymphoma;
23. T-cell lymphoma and NK/T-cell lymphoma with hemophagocytic syndrome;
24. Other situations deemed unsuitable for inclusion in the study by the researcher.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-12-31 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Best Objective Response Rate | On Day 1 of Cycle 4, Day 1 of Cycle 7, Day 1 of Cycle 10, Day 1 of Cycle 13, Day 1 of Cycle 16, Day 1 of Cycle 19, Day 1 of Cycle 22, and Day 1 of Cycle 25 (each cycle is 28 days)
  The rate of best overall response is the proportion of patients who achieve their best recorded response (complete or partial) to treatment at any time during the study.

SECONDARY OUTCOMES:
Complete remission rate | On Day 1 of Cycle 4, Day 1 of Cycle 7, Day 1 of Cycle 10, Day 1 of Cycle 13, Day 1 of Cycle 16, Day 1 of Cycle 19, Day 1 of Cycle 22, and Day 1 of Cycle 25 (each cycle is 28 days)
  Overall response rate is the proportion of patients who achieve a complete response to treatment defined by the Lugano classification criteria for lymphoma response evaluation (2014 edition).
Disease control rate | On Day 1 of Cycle 4, Day 1 of Cycle 7, Day 1 of Cycle 10, Day 1 of Cycle 13, Day 1 of Cycle 16, Day 1 of Cycle 19, Day 1 of Cycle 22, and Day 1 of Cycle 25 (each cycle is 28 days)
  Disease control rate is the proportion of patients who achieve either a complete or partial response to treatment defined by the Lugano classification criteria for lymphoma response evaluation (2014 edition).
Duration of Response | On Day 1 of Cycle 4, Day 1 of Cycle 7, Day 1 of Cycle 10, Day 1 of Cycle 13, Day 1 of Cycle 16, Day 1 of Cycle 19, Day 1 of Cycle 22, and Day 1 of Cycle 25 (each cycle is 28 days)
  Duration of response is the duration from the first documentation of a complete or partial response to disease progression or death.
Time To Response | On Day 1 of Cycle 4, Day 1 of Cycle 7, Day 1 of Cycle 10, Day 1 of Cycle 13, Day 1 of Cycle 16, Day 1 of Cycle 19, Day 1 of Cycle 22, and Day 1 of Cycle 25 (each cycle is 28 days)
  Time to response is the duration from the start of treatment to the first documentation of a complete or partial response.
Progression-free survival | From the first dose of treatment until the date of progression or date of death from any cause, whichever came first.
  PFS is defined as the time from the first dose of treatment to progression, or death due to any cause, whichever occurs first. For subjects without progression, relapse, or death at the time of analysis, EFS will be censored at the last assessment date.
Overall survival | From the first dose of treatment until the date of death from any cause
  OS is defined as the time from the first dose of treatment to death due to any cause. Subjects who remain alive at the time of analysis will be censored at the last known alive date of the subject.
Number of participants with any adverse events (Safety assessed by NCI-CTC AE v5.0) | Safety was evaluated everyday during induction and maintenance therapy. From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  All treatment-emergent AEs will be included in the analysis. For each AE, the number and percentage of subjects who experience at least one occurrence of the given event will be summarized. The number and percent of subjects with TEAEs will be summarized according to intensity (CTCAE, v5) for hematologic toxicity, and drug relationship, as well as categorized by system organ class and preferred term. Summaries, listings, datasets, or subject narratives may be provided, as appropriate, for those subjects who die, who discontinue treatment due to an AE, or who experience a severe AE or a SAE.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China